CLINICAL TRIAL: NCT03351101
Title: Clinical Study of Approved Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ROC2-17-014
Record Dates: First submitted 2017-11-09; First posted 2017-11-22 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: randomized, bilateral, d o u b l e - masked, 1-month study with two parallel groups
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Senofilcon C (Experimental): Senofilcon C Contact Lens
  Interventions: Device: Senofilcon C
- Samfilcon A (Experimental): Samfilcon A Contact Lens
  Interventions: Device: Samfilcon A

INTERVENTIONS:
Device: Senofilcon C — Senofilcon C Contact Lens
  Arms: Senofilcon C
Device: Samfilcon A — Samfilcon A Contact Lens
  Arms: Samfilcon A

SUMMARY:
Evaluation of Johnson & Johnson Acuvue Vita (senofilcon C) soft contact lenses to the Bausch + Lomb Ultra (samfilcon A) soft contact lenses

DETAILED DESCRIPTION:
to compare the performance of currently marketed Johnson & Johnson Acuvue Vita (senofilcon C) soft contact lenses to the currently marketed Bausch + Lomb Ultra (samfilcon A) soft contact lenses among adapted wearers of Acuvue Oasys soft contact lenses.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between the ages of 18 and 40 years old, inclusive, on the date the Informed Consent Form (ICF) is signed and have the capacity to provide voluntary informed consent.
2. Subjects must be able to read, understand and provide written informed consent on the Institutional Review Board (IRB)/Ethics Committee (EC) approved ICF and provide authorization as appropriate for local privacy regulations.
3. Subjects must be willing and able to comply with all treatment and follow-up/study procedures.
4. Subjects must be correctable through spherocylindrical refraction to 32 letters (0.3 logMAR) or better (distance, high contrast) in each eye.
5. Subjects must have clear central corneas and be free of any anterior segment disorders.
6. Subjects must be myopic and require contact lens sphere power correction from -0.50 diopter (D) to -6.00 D (considering vertex distance adjustments in both eyes).
7. Subjects must be habitual wearers of Johnson & Johnson Acuvue Oasys single vision spherical soft contact lenses in each eye.
8. Subjects must use a contact lens care regimen on a routine basis.
9. Subjects must agree to wear their study lenses on a daily wear basis for the duration

Exclusion Criteria:

1. Subjects participating in any drug or device clinical investigation within two weeks prior to entry into this study and/or during the period of study participation
2. Subjects who are women of childbearing potential (those who are not surgically sterilized or postmenopausal) are excluded from participation in the investigation if they meet any one of the following conditions:

   * she is currently pregnant
   * she plans to become pregnant during the study
   * she is breastfeeding
3. Subjects with any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an effect on ocular health during the course of the study.
4. Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - valeant Site 02, San Diego, California
  - Valeant Site 03, San Francisco, California
  - Valeant Site 04, Denver, Colorado
  - Valeant Site 06, Orlando, Florida
  - Valeant Site 01, Orlando, Florida
  - Valeant Site 05, Sarasota, Florida
  - Valeant Site 07, Pittsburg, Kansas
  - Valeant Site 08, Warrensburg, Missouri
  - Valeant Site 09, Vestal, New York
  - Valeant Site 10, Powell, Ohio
  - Valeant Site 11, New Berlin, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 271 participants enrolled, with 136 Senofilcon C participants dispensed lenses and 132 Samfilcon A participants dispensed lenses (268 participants total).
Period: Overall Study
Arm/Group | Senofilcon C | Samfilcon A
Started | 136 | 132
Completed | 135 | 129
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Population: All participants that completed all study visits without a major protocol deviation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Senofilcon C | Samfilcon A | Total
Number analyzed (Participants) | 115 | 106 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (5.62) | 30.4 (5.72) | 30.45 (5.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 68 | 139
  Male | 44 | 38 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 10 | 9 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 98 | 90 | 188
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: End of Day Comfort
Description: The 100 point , take home questionnaire evaluated performance of the lenses based on subject responses. Possible scores were 0-100. Higher scores indicated greater comfort.
Time Frame: 1 month
Population: All participants that completed all study visits without a major protocol deviation.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Senofilcon C | Samfilcon A
Number analyzed (Participants) | 115 | 106
score on a scale | 80 (18.15) | 80 (20.46)

2. Primary Outcome: Overall Vision
Description: The 100 point , take home questionnaire evaluated performance of the lenses based on subject responses. Possible scores were 0-100. Higher scores indicated better overall vision.
Time Frame: 1 month
Population: All participants that completed all study visits without a major protocol deviation.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Senofilcon C | Samfilcon A
Number analyzed (Participants) | 115 | 106
score on a scale | 95 (9.68) | 95 (12.15)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Senofilcon C | Samfilcon A
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/132
Other Adverse Events (participants affected / at risk) | 0/136 | 1/132
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Senofilcon C (N=136) | Samfilcon A (N=132)
Corneal infiltrates (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT03351101/Prot_SAP_000.pdf